CLINICAL TRIAL: NCT01499446
Title: A Randomised, Double-blind, Double Dummy, Placebo-controlled, Parallel-group Study to Evaluate the Efficacy and Safety of GW685698X 100mcg Administered Once Daily Either in the Morning or the Evening and GW685698X 250mcg Administered Once Daily in the Evening All Administered by Inhalation Via DISKHALER for 28 Days in Subjects With Persistent Bronchial Asthma.
Brief Title: A Study of GW685698X 100mcg Administered Once Daily Either in the Morning or the Evening and GW685698X 250mcg Administered Once Daily in the Evening Via DISKHALER for 28 Days in Subjects With Persistent Bronchial Asthma.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FFA20001
Record Dates: First submitted 2011-12-08; First posted 2011-12-26 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — fluticasone furoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- GW685698X (fluticasone furoate) 100mcg Morning (Experimental)
  Interventions: Drug: GW685698X (fluticasone furoate) 100mcg Morning
- GW685698X (fluticasone furoate) 100mcg Evening (Experimental)
  Interventions: Drug: GW685698X (fluticasone furoate) 100mcg Evening
- GW685698X (fluticasone furoate) 250mcg Evening (Experimental)
  Interventions: Drug: GW685698X (fluticasone furoate) 250mcg Evening
- Placebo (Placebo Comparator)
  Interventions: Drug: GW685698X (fluticasone furoate) 100mcg Morning; Drug: GW685698X (fluticasone furoate) 100mcg Evening; Drug: GW685698X (fluticasone furoate) 250mcg Evening; Drug: Placebo

INTERVENTIONS:
Drug: GW685698X (fluticasone furoate) 100mcg Morning — GW685698X inhaled once daily in the morning plus placebo in the evening for 28 days
  Arms: GW685698X (fluticasone furoate) 100mcg Morning; Placebo
Drug: GW685698X (fluticasone furoate) 100mcg Evening — GW685698X inhaled once daily in the evening fplus placebo in the morning for 28 days
  Arms: GW685698X (fluticasone furoate) 100mcg Evening; Placebo
Drug: GW685698X (fluticasone furoate) 250mcg Evening — GW685698X inhaled once daily in the evening plus placebo in the morning for 28 days
  Arms: GW685698X (fluticasone furoate) 250mcg Evening; Placebo
Drug: Placebo — Placebo inhaled twice daily (morning and evening) for 28 days
  Arms: Placebo

SUMMARY:
The purpose of this study is to compare the efficacy and safety of GW685698X 100mcg once daily either in the morning or the evening and GW685698X 250mcg administered once daily in the evening via DISKHALER for 28 days in subjects with persistent bronchial asthma.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients aged between 16- 65 years.
* Male and female; female subjects must be non-child bearing potential or of childbearing potenetial with negative pregnancy test and willing to use acceptable contraceptive methods
* Documented clinical history of persistent asthma first diagnosed at least 6 months prior to Visit 1
* Currently receiving inhaled short-acting beta-2 agonists for symptom relief
* A lung function of between 50 to 90% predicted (PEF)
* Increase in PEF of at least15%, 20 minutes after inhalation of 400mcg salbutamol

Exclusion Criteria:

* History of respiratory tract infection and/or exacerbation of asthma within a period of 4 weeks prior to Visit 1
* History of life-threatening asthma, defined as an asthma episode that required intubation and/or was associated with hypercapnoea, respiratory arrest or hypoxia seizures.
* A history of two or more asthma exacerbations requiring treatment with oral corticosteroids or hospitalisation in the 6 months before Visit 1.
* Past or present disease that, as judged by the investigator, may affect the outcome of this study. These diseases include, but are not limited to, cardiovascular disease, malignancy, hepatic disease, renal disease, haematologic disease, neurological disease, endocrine disease or pulmonary disease (including, but not confined to, chronic bronchitis, emphysema, bronchiectasis with the need of treatment, cystic fibrosis and bronchopulmonary dysplasia).
* Known or suspected sensitivity to corticosteroids, VENTOLIN, or the constituents of ROTADISKS (e.g., lactose).
* Undergoing allergen desensitisation therapy.
* Neurological or psychiatric disease or history of drug or alcohol abuse that would interfere with the subject's proper completion of the protocol requirements.
* Is a current smoker or has a smoking history of 10 pack years or more (e.g., 20 cigarettes/day for 10 years). Note: Current smoker is defined as currently smoking or stopped smoking within 6 months of screening visit.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 669 (Actual)
Dates: Start 2003-09; Primary Completion 2004-03 (Actual); Study Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
Peak expiratory flow (PEF) | 28 days
  Mean change from baseline in daily trough (pre study treatment and pre bronchodilator) PEF during the 28 day treatment period with GW685698X 100mcg once daily in the morning compared with GW685698X 100mcg once daily in the evening by inhalation via DISKHALER.

SECONDARY OUTCOMES:
Peak expiratory flow (PEF) | 28 days
  Mean change from baseline in daily trough (pre study treatment and pre bronchodilator) PEF during the 28 day treatment period with GW685698X 250mcg once daily compared with GW685698X 100mcg once daily both administered in the evening by inhalation via DISKHALER.
PEF | 28 days
  Mean change from baseline in daily trough (pre study treatment and pre bronchodilator) PEF during the 28 day treatment period with GW685698X 100mcg once daily in the morning, 100mcg once daily in the evening, or GW685698X 250mcg once daily in the evening, compared with placebo
Clinic lung function | 28 days
  Change from baseline in pre bronchodilator clinic lung function (forced expiratory volume in 1 second [FEV1] and PEF) after 28 days of treatment with GW685698X 250mcg once daily in the evening compared with GW685698X 100mcg once daily in the evening

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (50):
- GSK Investigational Site, Porto Alegre, Rio Grande do Sul, Brazil
- Bulgaria (3):
  - GSK Investigational Site, Pleven
  - GSK Investigational Site, Sofia
  - GSK Investigational Site, Varna
- GSK Investigational Site, Santiago, Región Metro de Santiago, Chile
- Croatia (3):
  - GSK Investigational Site, Osijek
  - GSK Investigational Site, Split
  - GSK Investigational Site, Zagreb
- Estonia (4):
  - GSK Investigational Site, Kohtal-Jdrve
  - GSK Investigational Site, Pärnu
  - GSK Investigational Site, Tallinn
  - GSK Investigational Site, Tartu
- Germany (13):
  - GSK Investigational Site, Schwetzingen, Baden-Wurttemberg
  - GSK Investigational Site, Weinheim, Baden-Wurttemberg
  - GSK Investigational Site, Eschwege, Hesse
  - GSK Investigational Site, Gelnhausen, Hesse
  - GSK Investigational Site, Kassel, Hesse
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Lüneburg, Lower Saxony
  - GSK Investigational Site, Gütersloh, North Rhine-Westphalia
  - GSK Investigational Site, Annaberg, Saxony
  - GSK Investigational Site, Aue, Saxony
  - GSK Investigational Site, Geesthacht, Schleswig-Holstein
  - GSK Investigational Site, Berlin, State of Berlin
  - GSK Investigational Site, Erfurt, Thuringia
- Greece (2):
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Papagos/Athens
- GSK Investigational Site, Törökbálint, Hungary
- Italy (11):
  - GSK Investigational Site, Eboli (SA), Campania
  - GSK Investigational Site, Napoli, Campania
  - GSK Investigational Site, Salerno, Campania
  - GSK Investigational Site, Ferrara, Emilia-Romagna
  - GSK Investigational Site, Genoa, Liguria
  - GSK Investigational Site, Sesto San Giovanni (MI), Lombardy
  - GSK Investigational Site, Torrette (AN), The Marches
  - GSK Investigational Site, Florence, Tuscany
  - GSK Investigational Site, Pisa, Tuscany
  - GSK Investigational Site, Bussolengo (VR), Veneto
  - GSK Investigational Site, Padua, Veneto
- Mexico (2):
  - GSK Investigational Site, Mexico City
  - GSK Investigational Site, México
- Romania (2):
  - GSK Investigational Site, Brasov
  - GSK Investigational Site, Bucharest
- Russia (5):
  - GSK Investigational Site, Kazan'
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Tomsk
  - GSK Investigational Site, Volgograd
- South Africa (2):
  - GSK Investigational Site, Bloemfontein
  - GSK Investigational Site, Cape Town

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] O'Byrne PM, Jacques L, Goldfrad C, Kwon N, Perrio M, Yates LJ, Busse WW. Integrated safety and efficacy analysis of once-daily fluticasone furoate for the treatment of asthma. Respir Res. 2016 Nov 24;17(1):157. doi: 10.1186/s12931-016-0473-x. PMID 27881132
- [Derived] Medley H, Orozco S, Allen A. Efficacy and safety profile of fluticasone furoate administered once daily in the morning or evening: a randomized, double-blind, double-dummy, placebo-controlled trial in adult and adolescent patients with persistent bronchial asthma. Clin Ther. 2012 Aug;34(8):1683-95. doi: 10.1016/j.clinthera.2012.06.024. Epub 2012 Jul 13. PMID 22796247
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: FFA20001 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: FFA20001 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: FFA20001 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: FFA20001 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: FFA20001 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: FFA20001 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: FFA20001 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register